CLINICAL TRIAL: NCT03641352
Title: The Efficacy and Safety of CKD-501 Added to D150 Plus D759 Therapy in Patients With Type 2 Diabetes Inadequately Controlled With D150 Plus D759, Randomized, Double-blind, Multi-center, Parallel-group, Placebo Control, Therapeutic Confirmatory Study
Brief Title: The Efficacy and Safety of CKD-501 Added to D150 Plus D759 Therapy in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19DM17012
Record Dates: First submitted 2018-07-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-501 0.5mg (Experimental): CKD-501 0.5mg
  Interventions: Drug: CKD-501 0.5mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-501 0.5mg — CKD-501 0.5mg, orally, 1 tablet once a dqy for 24weeks or 52weeks (if extension study) with D150 and D759
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: Placebo — Placebo, orally, 1 tablet once a dqy for 24weeks or 52weeks (if extension study) with D150 and D759. CKD-501 placebo will be changed to CKD-501 from extension study to EOS(end of study).
  Arms: Placebo

SUMMARY:
The purpose of this study is to prove that the group treated with CKD-501 in combination added that the reduction of glycated hemoglobin superior to placebo treated group added in combination.

DETAILED DESCRIPTION:
The aim of this phase 3 study was to evaluate the efficacy and safety of additional combined CKD-501 administration for 24 weeks in patient with type 2 diabetes who were nao adequately controlled for blood glucose by the combination of D150 and D759

ELIGIBILITY:
Inclusion Criteria:

* between 19 years and 80 years old(male or female)
* Type 2 diabetes mellitus
* The patient who has been taking oral hypoglycemic agent at least 8weeks with HbA1c 7 to 10% at screening test
* BMI between 21kg/m2 and 40kg/m2
* C-peptide ≥ 1.0 ng/ml
* Agreement with written informed consent
* HbA1c 7 to 10% after Run-in period

Exclusion Criteria:

* Type 1 diabetes mellitus or secondary diabetes mellitus
* Continuous or non continuous treatment(over 7 days) insulin within 3 months prior to screening
* Treatment with Thiazolidinedione(TZD) within 3 months or patient who has experience such as hypersensitivity reaction, serious adverse event with TZD, Biguanide
* Chronic(continuous over 7 days) oral or non oral corticosteroids treatment within 1 month prior to screening
* Treatment with anti-obesity drugs within 3 months

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin | Baseline, 24weeks

SECONDARY OUTCOMES:
Change from baseline in in Glycosylated Hemoglobin | Baseline, 52weekes
Change from baseline in Fasting plasma glucose | Baseline, 24weeks, 52weeks
HbA1c target achievement rate at 24weekes(HbA1c < 6.5%, 7%) | Baseline, 24weeks
Change from baseline in Total Cholesterol | Baseline, 24weeks, 52weeks
Evaluate safety of CKD-501 from number of participants with adverse events | Baseline, 24weeks, 52weeks
Change from baseline in HOMA-IR(Homeostasis Model Assessment of Insulin Resistance) | Baseline, 24weeks, 52weeks
Change from baseline in HOMA-β(Homeostasis Model Assessment of β-cell function) | Baseline, 24 weeks, 52 weeks
Change from baseline in QUICKI(Quantitative Insulin Check Index) | Baseline, 24 weeks, 52 weeks
Change from baseline in Triglycerides | Baseline, 24 weeks, 52 weeks
Change from baseline in LDL-Cholesterol | Baseline, 24 weeks, 52 weeks
Change from baseline in HDL-Cholesterol | Baseline, 24 weeks, 52 weeks
Change from baseline in non-HDL-Cholesterol | Baseline, 24 weeks, 52 weeks
Change from baseline in Small Dense LDL-Cholesterol | Baseline, 24 weeks, 52 weeks
Change from baseline in FFA(Free Fatty Acid) | Baseline, 24 weeks, 52 weeks
Change from baseline in Apo-B | Baseline, 24 weeks, 52 weeks
Change from baseline in Apo-CⅢ | Baseline, 24 weeks, 52 weeks
Change from baseline in Apo-AⅠ | Baseline, 24 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kun ho Yoon, Ph.D, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No